CLINICAL TRIAL: NCT07391033
Title: Impact of Lesion PREParation With Modifying Balloons During Drug-coated Balloon (DCB) Angioplasty for In-stent Restenosis (ISR) - PICCOLETO XI A-PREP Study
Brief Title: The PICCOLETO XI A-PREP Study
Acronym: PICCOLETO-XI
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Ricerca e Innovazione Cardiovascolare ETS (Other)
Responsible Party: Sponsor
Other Study IDs: PICCOLETO XI
Record Dates: First submitted 2026-01-29; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: In-Stent Coronary Artery Restenosis; Coronary Artery Disease
Keywords: Drug-Coated Balloon; In-Stent Restenosis; Lesion Preparation; Cutting Balloon; Scoring Balloon; Percutaneous Coronary Intervention
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Aggressive Lesion Preparation: Patients who underwent lesion preparation using cutting/Wolverine balloons, scoring balloons (any brand), and/or OPN balloons prior to DCB angioplasty for ISR.
- Standard Lesion Preparation: Patients who underwent lesion preparation using semi-compliant balloons and/or non-compliant balloons prior to DCB angioplasty for ISR.

SUMMARY:
To compare the angiographic and clinical outcomes of aggressive versus standard balloon preparation during drug-coated balloon (DCB) angioplasty for in-stent restenosis (ISR). The study will evaluate whether more aggressive lesion preparation with cutting/scoring/OPN balloons improves outcomes compared to standard preparation with semi-compliant or non-compliant balloons.

DETAILED DESCRIPTION:
PICCOLETO XI A-PREP is an investigator-initiated, multicenter, international, observational study evaluating the impact of lesion preparation strategies on outcomes following drug-coated balloon (DCB) angioplasty for in-stent restenosis (ISR).

In-stent restenosis remains a clinically relevant challenge despite advances in drug-eluting stent technology and contemporary percutaneous coronary intervention techniques. DCB represents a stentless therapeutic strategy for ISR treatment, with the advantage of avoiding implantation of additional metallic layers.

A key determinant of clinical outcomes in ISR, particularly with DCB angioplasty, is the adequacy of lesion preparation before definitive therapy. Effective preparation facilitates optimal drug delivery, improves luminal gain, and may reduce the risk of recurrent restenosis.

A large spectrum of balloon-based modalities is available for ISR lesion preparation, ranging from semi-compliant and non-compliant balloons to more aggressive tools such as scoring and cutting balloons. Although more aggressive devices may enhance plaque modification and neointimal tissue disruption, their incremental clinical benefit over standard approaches remains uncertain.

Patients will be categorized into two groups based on lesion preparation strategy:

* Aggressive preparation: Cutting/Wolverine balloons, scoring balloons (any brand), and/or OPN balloons
* Standard preparation: Semi-compliant balloons and/or non-compliant balloons

Clinical outcomes will be assessed at 1-year and longest available follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥18 years of age
* Patients who underwent DCB angioplasty for in-stent restenosis

Exclusion Criteria:

- Lack of clinical outcome assessment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who underwent drug-coated balloon (DCB) angioplasty for in-stent restenosis (ISR) at participating centers.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiovascular Events (MACE) | 12 months
  Composite of cardiac death, non-fatal myocardial infarction (MI), or target lesion revascularization (TLR).

SECONDARY OUTCOMES:
Cardiac Death | 12 months and longest available follow-up
  Death attributed to cardiovascular causes, including death from unknown cause.
Non-fatal Myocardial Infarction | 12 months and longest available follow-up
  Non-fatal myocardial infarction according to the Fourth Universal Definition of Myocardial Infarction.
Target Lesion Revascularization (TLR) | 12 months and longest available follow-up
  Any repeat revascularization (percutaneous or surgical) of the target lesion.
Target Vessel Myocardial Infarction (TV-MI) | 12 months and longest available follow-up
  Myocardial infarction attributable to the target vessel based on clinical, electrocardiographic, and biomarker criteria.
BARC Major Bleeding | 12 months and longest available follow-up
  Bleeding Academic Research Consortium (BARC) major bleeding events (type 3-5).
Procedural Success | At procedure
  Successful DCB angioplasty with residual stenosis less than 30% and TIMI flow grade 3 without major procedural complications.
Post-procedural Diameter Stenosis | At procedure
  Percentage of diameter stenosis after DCB angioplasty assessed by quantitative coronary angiography.
Angiographic Dissection | At procedure
  Presence and type of coronary dissection after lesion preparation and DCB treatment.
TIMI Flow Grade | At procedure
  Thrombolysis In Myocardial Infarction (TIMI) flow grade assessment post-procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Bharat Khialani, MD, Principal Investigator — Tan Tock Seng Hospital, National Healthcare Group, Singapore; Filippo Luca Gurgoglione, MD, PhD, Principal Investigator — Department of Cardiology, Parma University Hospital, Parma, Italy; Bernardo Cortese, MD, Study Chair — Fondazione Ricerca e Innovazione Cardiovascolare ETS

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data may be made available to qualified researchers upon reasonable request after study completion and primary publication, subject to appropriate data use agreements and ethics committee approval.

REFERENCES:
- [Background] Wańha W, Iwańczyk S, Tajstra M, Cortese B. How to treat coronary in-stent restenosis? Recent advances and their practical implications: State-of-the-Art Review. Kardiol Pol. 2025;83(5):556-569. doi: 10.33963/v.phj.105954.
- [Background] Dangas GD, Claessen BE, Caixeta A, Sanidas EA, Mintz GS, Mehran R. In-stent restenosis in the drug-eluting stent era. J Am Coll Cardiol. 2010;56:1897-907. doi: 10.1016/j.jacc.2010.07.028.
- [Background] Latib A, Mussardo M, Ielasi A, Tarsia G, Godino C, Al-Lamee R, Chieffo A, Airoldi F, Carlino M, Montorfano M, Colombo A. Long-term outcomes after the percutaneous treatment of drug-eluting stent restenosis. JACC Cardiovasc Interv. 2011;4:155-64. doi: 10.1016/j.jcin.2010.09.027.
- [Background] Mauri L, Bonan R, Weiner BH, et al. Cutting balloon angioplasty for the prevention of restenosis: results of the Cutting Balloon Global Randomized Trial. Am J Cardiol. 2002;90(10):1079-1083. doi: 10.1016/S0002-9149(02)02773-X.
- [Background] Bonaventura K, Schwefer M, Yusof AKM, Waliszewski M, Krackhardt F, Steen P, Ocaranza R, Zuhdi AS, Bang LH, Graf K, Böck U, Chin K. Systematic Scoring Balloon Lesion Preparation for Drug-Coated Balloon Angioplasty in Clinical Routine: Results of the PASSWORD Observational Study. Adv Ther. 2020 May;37(5):2210-2223. doi: 10.1007/s12325-020-01320-2.